CLINICAL TRIAL: NCT00109980
Title: Dominican Herbal Medicine: Plants Used for Inflammation
Brief Title: Medicinal Plant Use for Treating Inflammation Among Dominicans in New York City and the Dominican Republic
Status: Completed | Type: Observational
Sponsor: New York Botanical Garden (Other)
Responsible Party: Principal Investigator, Michael Balick, Director, National Center for Complementary and Integrative Health (NCCIH)
Other Study IDs: R21AT001889-01A1 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Inflammation
Keywords: Complementary Therapies; Plants, Medicinal; Dominican Republic; Hispanic Americans
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate and compare the use of herbal medicine among Dominicans in New York City and the Dominican Republic.

DETAILED DESCRIPTION:
According to the 2000 U.S. Census Report, Dominicans constitute the largest Hispanic immigrant group in New York City. Studies have shown that immigrants' use of traditional and herbal medicine is close to that of native-born Americans. However, minority immigrants often have limited access to traditional health care; as a result, they may be more likely to consult with traditional healers and use medicinal plants than nonimmigrants. This study is designed to increase knowledge about immigrants' health and to contribute to more culturally-sensitive health care. The purpose of this study is to determine medical plant knowledge and use among Dominican traditional healers and patients in New York City and in the Dominican Republic.

This study will comprise two parts. In Part I, Dominican medicinal plant users and Dominican traditional healers in New York City will be questioned about the medicinal plant species they know and how they are used for prevalent illnesses. The same number of participants will be interviewed in the Dominican Republic, allowing for detailed comparisons between the two study sites.

In Part II, the most frequently-cited medicinal plant species will be subjected to a thorough literature review on their pharmacologic activity and the chemical composition of their active constituents. Two in vitro assays will be used to measure the anti-inflammatory activity of certain plant extracts, and their anti-inflammatory compounds will be isolated and characterized for the purpose of standardization of active extracts. On the basis of these results, recommendations will be formulated for future studies and community use of selected medicinal plant species.

ELIGIBILITY:
Inclusion Criteria:

* Dominican ethnicity
* Have knowledge of Dominican medicinal plants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dominican community sample in New York City
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2005-03; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Identification of culturally important medicinal plants | June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Balick, PhD, Principal Investigator — Institute of Economic Botany, the New York Botanical Garden
Locations (1):
- Associates in Internal Medicine Clinic, New York-Presbyterian Hospital, Columbia University, New York, New York, United States

REFERENCES:
- [Background] Balick MJ, Kronenberg F, Ososki AL, Reiff M, Fugh-Berman A, O'Connor B, Roble M, Lohr P, Atha D. Medicinal plants used by Latino healers for women's health conditions in New York City. Economic Botany 54: 344-357, 2000.
- [Background] Balick MJ, Lee R. Looking within: urban ethnomedicine and ethnobotany. Altern Ther Health Med. 2001 Jul-Aug;7(4):114-5. No abstract available. PMID 11452554
- [Background] Fugh-Berman A, Balick MJ, Kronenberg F, Ososki AL, O'Connor B, Reiff M, Roble M, Lohr P, Brosi BJ, Lee R. Treatment of fibroids: the use of beets (Beta vulgaris) and molasses (Saccharum officinarum) as an herbal therapy by Dominican healers in New York City. J Ethnopharmacol. 2004 Jun;92(2-3):337-9. doi: 10.1016/j.jep.2004.03.009. No abstract available. PMID 15138021
- [Background] Ososki AL, Lohr P, Reiff M, Balick MJ, Kronenberg F, Fugh-Berman A, O'Connor B. Ethnobotanical literature survey of medicinal plants in the Dominican Republic used for women's health conditions. J Ethnopharmacol. 2002 Mar;79(3):285-98. doi: 10.1016/s0378-8741(01)00376-2. PMID 11849831
- [Background] Reiff M, O'Connor B, Kronenberg F, Balick M, Lohr P, Roble M, Fugh-Berman A, Johnson KD. Ethnomedicine in the urban environment: Dominican healers in New york City. Human Organization 62(1): 12-26, 2003.
- [Background] Vandebroek I, Balick MJ, Yukes J, Duran L, Kronenberg F, Wade C, Ososki AL, Cushman L, Lantigua R, Mejia M & Robineau L (2007) Use of medicinal plants by Dominican immigrants in New York City for the treatment of common health conditions. A comparative analysis with literature data from the Dominican Republic. In: A. Pieroni & I. Vandebroek, eds., Traveling Cultures and Plants: The Ethnobiology and Ethnopharmacy of Human Migrations. Bergahn Books, New York, pp. 39-63.